CLINICAL TRIAL: NCT00220519
Title: Lactobacillus GG Supplementation During Pediatric Burn Injuries
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped due to low enrollment
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Maggie L. Dylewski, Shriners Hospitals for Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2004-P-001990/1
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2005-09

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lactobacillus GG

SUMMARY:
Critical illness and the therapies that accompany it are associated with a disruption in the ecological equilibrium of the GI tract that can ultimately lead to infection. Lactobacillus GG, a probiotic, replenishes the healthy flora of the intestinal tract and may decrease the risk of diarrhea and infection during critical illness. However, little is known about the impact of probiotics following a burn injury and the mechanisms behind the proposed benefits. The hypothesis of this research is that Lactobacillus GG decreases the incidence of diarrhea and infection in burned children receiving antibiotic therapy. The specific aim of this research is to determine the impact of Lactobacillus GG on the incidence of diarrhea and infection among burned children (>20% TBSA) receiving antibiotic therapy.

DETAILED DESCRIPTION:
Specific Aim:

Critical illness and the therapies that accompany it are associated with a disruption in the ecological equilibrium of the GI tract that can ultimately lead to infection. Lactobacillus GG, a probiotic, repletes the healthy flora of the intestinal tract and may decrease the risk of diarrhea and infection during critical illness. However, little is known about the impact of probiotics following a burn injury and the mechanisms behind the proposed benefits. The hypothesis of this research is that Lactobacillus GG decreases the incidence of diarrhea and infection in burned children receiving antibiotic therapy. The specific aim of this research is to determine the impact of Lactobacillus GG on the incidence of diarrhea and infection among burned children (>20% TBSA) receiving antibiotic therapy.

Subjects:

All subjects will be recruited from the Shriners Hospitals for Children in Boston. Patients of any age admitted to Shriners Hospitals for Children in Boston that match the following inclusion criteria will be considered for this study 1)burn wound size of at least 20% of the body surface area, 2)requires antibiotic therapy. Exclusion criteria includes: 1) < 20% total body surface area burn, 2)does not require antibiotic therapy, 3)only requires post-operative antibiotic therapy, 4)bowel obstruction, 5)milk allergy.

Study Design:

This is a randomized, double-blind, placebo-controlled trial. Patients will be randomly assigned to receive Lactobacillus GG (n = 47) or a placebo (n = 47) within 3 days of initiation of antibiotic therapy. Randomization will occur by using a computerized randomization list. A pharmacist, who is not a member of the study staff, will assign each of the 2 supplement groups a number and label the supplement bottles accordingly.

Methods:

Lactobacillus GG, a nonpathogenic microorganism, will be administered in this study. A dose of 1010 colony factor units (cfu) twice daily will be given to the experimental group (n =47). The control group will receive a placebo (n = 47) that will be identical in appearance to the probiotic. All supplements will be administered orally or via feeding tube. The study endpoint will be 10 days after antibiotic use is discontinued or patient discharge Parameters measured will include 1) the occurrence of pneumonia or infection in the wound, blood, or urine, as defined by The National Nosocomial Infection Surveillance System (A localized or systemic condition that results from adverse reaction to the presence of an infectious agent(s) or toxin(s)) and clarified by the Infection Control Nurse, 2) incidence of diarrhea defined as 3 or more loose or watery stools per 24 hours, 3) weekly weights and labs (including total protein, albumin, prealbumin and C-reactive protein) as obtained per routine care, 4) length of antibiotic use, 5) length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Burn wound size of at least 20% of the body surface area
* Requires antibiotic therapy

Exclusion Criteria:

* < 20% total body surface area burn
* Does not require antibiotic therapy
* Only requires post-operative antibiotic therapy
* Bowel obstruction
* Milk allergy

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2004-10; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Infection | Daily
Diarrhea | Daily

CONTACTS AND LOCATIONS:
Overall Officials: Maggie L Dylewski, MS,RD, Principal Investigator — Shriners Hospitals for Children
Locations (1):
- Shriners Hospitals for Children, Boston, Massachusetts, United States